CLINICAL TRIAL: NCT05488730
Title: Role of Echocardiography in Guiding Fluid Therapy in Shocked Patients With Impaired Cardiac Contractility in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mostafa Gaber, assistant lecturer of emergency medicine, Alexandria University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Echo in fluid therapy 2022
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- shocked patient with impaired cardiac contractility (Other)
  Interventions: Diagnostic Test: passive leg raising test and fluid challenge

INTERVENTIONS:
Diagnostic Test: passive leg raising test and fluid challenge — Shocked patients were subjected to echocardiographic examination if (EF <52%) .baseline LVOT VTI was obtained Then IVC scanning was done through subcostal Window and using M-mode the minimum and the maximum diameters were measured then the collapsibility index was calculated
  Then passive leg raising test was done Patients who tolerated the PLR test and did not develop clinical or lung ultrasound signs of fluid overload (lung congestion) were given IV fluid bolus (250 ml normal saline) over 10 minutes followed by measurement of LVOT VTI.
  Patients who did not tolerate PLR test or developed clinical or lung ultrasound signs of fluid overload (lung congestion) during PLR test were excluded from the third step (fluid challenge).
  The differentiating factor used to allocate patient in which group (non-responder or responder) was LVOT VTI variability after fluid challenge (our gold standard to assess fluid responsiveness).

SUMMARY:
fluid therapy is one of the cornerstones in the management of shock but may result in iatrogenic fluid overload .The aim of this study was to assess the role of echocardiography in guiding fluid therapy in shocked patients with impaired cardiac contractility using straight leg raising test ,Inferior vena-cava collapsability index and Doppler imaging in Emergency Department in Alexandria main university hospital.

ELIGIBILITY:
Inclusion Criteria:

* shocked patient with impaired cardiac contractility

Exclusion Criteria:

* Trauma patients.
* Patient with unstable arrhythmias.
* Patients with lower limb amputation.
* Mechanically ventilated patients.
* Patients with prosthetic aortic valve.
* Patients less than 18 years old
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
LVOT VTI variability | 15 minutes
  variability of LVOT VTI to determine fluid responsiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
study protocol to be shared later after publishing my scientific paper